CLINICAL TRIAL: NCT00177840
Title: Acupuncture for Cancer-Related Fatigue in Breast Cancer Patients
Brief Title: Acupuncture to Treat Cancer-Related Fatigue in Breast Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Judith Balk, University of Pittsburgh
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 0506139; R21CA098659-01A2 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Fatigue
Keywords: cancer-related fatigue; acupuncture; breast cancer
MeSH Terms: conditions — Fatigue; Breast Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): True acupuncture using true needles
  Interventions: Procedure: acupuncture
- 2 (Sham Comparator): sham acupuncture using sham needles
  Interventions: Procedure: acupuncture

INTERVENTIONS:
Procedure: acupuncture

SUMMARY:
This study will evaluate if acupuncture is helpful in treating cancer-related fatigue in breast cancer patients undergoing radiation therapy.

DETAILED DESCRIPTION:
Each participant will have a baseline visit before her radiation therapy begins to complete questionnaires. Participants will receive either true acupuncture or sham acupuncture twice per week for the six weeks of radiation therapy. She will have a short questionnaire at three weeks into her radiation, and she will complete questionnaires again at the end of her radiation and four weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Localized breast cancer
* Average to above average fatigue
* Planning radiation therapy

Exclusion Criteria:

* History of acupuncture treatment
* Allergy to stainless steel
* Pacemaker
* Anticoagulant therapy
* Known bleeding disorder
* Metastatic breast cancer
* Seizure disorder

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2005-09; Primary Completion 2007-07 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Cancer-related fatigue | 10 weeks

SECONDARY OUTCOMES:
Cancer-related fatigue distress | 10 weeks
Quality of life | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Judith Balk, MD MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States